CLINICAL TRIAL: NCT00996138
Title: A Multi-center, Randomized, Single-blind, Dose-Ranging Study to Evaluate Immunogenicity, Safety and Tolerability of Different Doses of Adjuvanted Cell-Derived, Inactivated Novel Swine Origin A/H1N1 Monovalent Subunit Influenza Virus Vaccine in Healthy Japanese Adult Subjects
Brief Title: Single-blind, Dose-ranging Study of Novel Swine Influenza Virus Vaccine in Japanese Adult Subjects
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V110_05
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2012-09

CONDITIONS: Influenza
Keywords: Influenza A; H1N1 subtype; Adult; Vaccine; Adjuvant; Swine-Origin Influenza A H1N1 Virus
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Arm 1 (Other): Dose ranging
  Interventions: Biological: Adjuvanted cell-derived, inactivated novel swine origin A/H1N1 monovalent subunit influenza virus vaccine
- Arm 2 (Other): Dose ranging
  Interventions: Biological: Adjuvanted cell-derived, inactivated novel swine origin A/H1N1 monovalent subunit influenza virus vaccine

INTERVENTIONS:
Biological: Adjuvanted cell-derived, inactivated novel swine origin A/H1N1 monovalent subunit influenza virus vaccine — High dose group and low dose group of adjuvanted vaccines

SUMMARY:
This study is to identify the preferred vaccine dosage (of antigen and adjuvant) and schedule (one or two administrations) of the cell-derived H1N1sw monovalent vaccine in healthy adults based on EMEA/CHMP criteria, and safety & tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese adults aged 20 to 60 years

Exclusion Criteria:

* History of anaphylaxis, serious vaccine reactions, hypersensitivity to vaccine viral proteins or excipients
* Administration of adjuvanted influenza vaccine or suspected influenza disease within 3 month prior to study start
* Administration of any other vaccines within 4 weeks prior to enrollment expect for seasonal influenza vaccines within 1 week
* History of progressive or severe neurological disorders

Ages: 29 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Seroprotection, GMRs and Seroconversion rate at Weeks 0, 3 and 6 | 6 weeks

SECONDARY OUTCOMES:
AEs, vital signs, laboratory tests | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Osaka pref., Kagoshima Pref., Japan

REFERENCES:
- [Result] Fukase H, Furuie H, Yasuda Y, Komatsu R, Matsushita K, Minami T, Suehiro Y, Yotsuyanagi H, Kusadokoro H, Sawata H, Nakura N, Lattanzi M. Assessment of the immunogenicity and safety of varying doses of an MF59(R)-adjuvanted cell culture-derived A/H1N1 pandemic influenza vaccine in Japanese paediatric, adult and elderly subjects. Vaccine. 2012 Jul 13;30(33):5030-7. doi: 10.1016/j.vaccine.2012.03.053. Epub 2012 Apr 1. PMID 22472791